CLINICAL TRIAL: NCT02571972
Title: Effect of Topical Aqueous Suppressants on Response to Intravitreal Anti-vascular Endothelial Growth Factor Injections in Age-related Macular Degeneration (AMD), Retinal Vein Occlusions (RVO) or Diabetic Macular Edema (DME).
Brief Title: Dorzolamide-timolol Drops With Injections to Treat AMD, RVO or DME.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: J. Arch McNamara Research Fund (Other); Mid Atlantic Retina (Other)
Responsible Party: Principal Investigator, Jason Hsu, MD, PI, Wills Eye
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#14-435
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Wet Macular Degeneration; Age-related Macular Degeneration; Diabetic Macular Edema; Retinal Vein Occlusion
Keywords: dorzolamide-timolol; topical aqueous suppression; neovascular age-related macular degeneration; macular edema; intravitreal injection; anti-vascular endothelial growth factor
MeSH Terms: conditions — Wet Macular Degeneration; Macular Degeneration; Retinal Vein Occlusion; Macular Edema | interventions — dorzolamide-timolol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dorzolamide-timolol (Experimental): * On enrollment, eligible patients will have visual acuity testing, intraocular pressure, dilated fundoscopic examination, SD-OCT scan and will then receive the same intravitreal pharmacologic agent administered at prior visit.
  * Subsequent follow-up visits will be at an identical interval to pre-enrollment visit intervals (4, 5, or 6 week intervals) for the study duration.
  * Each subsequent visit will consist of visual acuity testing, intraocular pressure, dilated fundoscopic examination, SD-OCT scan, and intravitreal injection of same pharmacologic agent as prior visits
  * At study conclusion, mean central macular thickness, maximum subretinal fluid height, and maximum pigment epithelial detachment height will be measured over the study period for all patients
  Interventions: Drug: Dorzolamide-timolol

INTERVENTIONS:
Drug: Dorzolamide-timolol — On enrollment, eligible patients will be started on topical dorzolamide-timolol in the study eye twice daily for the study duration
  Other Names: Cosopt

SUMMARY:
This study seeks to evaluate the effect of topical aqueous suppression on the anatomic and functional response to intravitreal anti-vascular endothelial growth factor (VEGF) injections in non-responders with wet age-related macular degeneration.

DETAILED DESCRIPTION:
Intravitreal anti-vascular endothelial growth factor (VEGF) agents, including bevacizumab, ranibizumab, and aflibercept, have become the gold standard treatment for neovascular age-related macular degeneration (AMD). Various treatment modalities using these agents have been proposed, including monthly, pro re nata, and treat-and-extend philosophies. Despite frequent and consistent treatment with anti-VEGF therapy, there is a subset of patients who are incomplete or non-responders and have persistent evidence of exudation on spectral-domain optical coherence tomography (SD-OCT), including subretinal fluid (SRF) and/or intraretinal edema.

While clearance of intravitreal anti-VEGF drugs is not completely understood, some studies have suggested that outflow through the anterior chamber may contribute. We hypothesized that by decreasing aqueous production, outflow may also be reduced which could delay the clearance of intravitreal drugs. As a result, we chose topical dorzolamide-timolol since it is a potent aqueous suppressant and is readily available due to its common use in the treatment of glaucoma. The current study aimed to evaluate the efficacy of topical dorzolamide-timolol on anatomic and visual outcomes in anti-VEGF non-responders with neovascular AMD.

Significance: The results of this study will help delineate whether topical aqueous suppression may be useful as adjuvant therapy in patients receiving chronic intravitreal anti-VEGF injections.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of Wills Eye Hospital Retina Service and/or Mid Atlantic Retina.
2. Volunteer patients age 18 years and older.
3. Healthy enough to participate in the study.
4. Willing and able to consent to participation in the study.
5. Diagnosis of wet age-related macular degeneration
6. Prior treatment with at least 4 injections of anti-VEGF agents in the past 6 months and persistent intraretinal and/or subretinal fluid on SD-OCT at each visit during this period
7. Injection of the same anti-VEGF agent for at least two visits prior to study enrollment
8. Fixed interval between at least two visits prior to study enrollment

Exclusion Criteria:

1. History of uveitis
2. Any ophthalmic surgery within previous 6 months, including cataract extraction.
3. Any history of vitrectomy
4. History of any glaucoma drop usage or prior glaucoma surgery
5. Systemic diuretic or corticosteroid usage
6. Any contraindication (bradycardia, decompensated heart failure, or reactive
7. airway disease) for topical use of a beta-blocker
8. Any history of sulfonamide allergy

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hsu, MD, Principal Investigator — Wills Eye Hospital, Mid Atlantic Retina
Locations (1):
- Wills Eye Hospital / Mid Atlantic Retina, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byeon SH, Kwon OW, Song JH, Kim SE, Park YS. Prolongation of activity of single intravitreal bevacizumab by adjuvant topical aqueous depressant (Timolol-Dorzolamide). Graefes Arch Clin Exp Ophthalmol. 2009 Jan;247(1):35-42. doi: 10.1007/s00417-008-0917-1. Epub 2008 Aug 6. PMID 18682969
- [Result] Sridhar J, Hsu J, Shahlaee A, Garg SJ, Spirn MJ, Fineman MS, Vander J. Topical Dorzolamide-Timolol With Intravitreous Anti-Vascular Endothelial Growth Factor for Neovascular Age-Related Macular Degeneration. JAMA Ophthalmol. 2016 Apr;134(4):437-43. doi: 10.1001/jamaophthalmol.2016.0045. PMID 26914218
- [Derived] Obeid A, Hsu J, Ehmann D, Gao X, Sridhar J, Chiang A, Park CH, Ho AC. TOPICAL DORZOLAMIDE-TIMOLOL WITH INTRAVITREOUS ANTI-VASCULAR ENDOTHELIAL GROWTH FACTOR FOR RETINAL VEIN OCCLUSION: A PILOT STUDY. Retin Cases Brief Rep. 2021 Mar 1;15(2):120-126. doi: 10.1097/ICB.0000000000000752. PMID 29864044

RESULTS

PARTICIPANT FLOW:
Groups:
- Dorzolamide-timolol: On enrollment, eligible patients will be started on topical dorzolamide 2%-timolol 0.5% 1 drop in the study eye twice daily for the study duration
Period: Overall Study
Arm/Group | Dorzolamide-timolol
Started | 14 (2 patients signed consent but withdrew from the study prior to using dorzolamide-timolol drops.)
Completed | 10
Not Completed | 4
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Dorzolamide-timolol: * On enrollment, eligible patients will have visual acuity testing, intraocular pressure, dilated fundoscopic examination, SD-OCT scan and will then receive the same intravitreal pharmacologic agent administered at prior visit.
  * Subsequent follow-up visits will be at an identical interval to pre-enrollment visit intervals (4, 5, or 6 week intervals) for the study duration.
  * Each subsequent visit will consist of visual acuity testing, intraocular pressure, dilated fundoscopic examination, SD-OCT scan, and intravitreal injection of same pharmacologic agent as prior visits
  * At study conclusion, mean central macular thickness, maximum subretinal fluid height, and maximum pigment epithelial detachment height will be measured over the study period for all patients
  Dorzolamide-timolol: On enrollment, eligible patients will be started on topical dorzolamide-timolol in the study eye twice daily for the study duration
Arm/Group | Dorzolamide-timolol
Number analyzed (Participants) | 10
Number analyzed (Eyes) | 10
Age, Continuous [Mean (Full Range); unit: years] | 78.2 [65 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Intravitreous anti-vascular endothelial growth factor (VEGF) agent [Count of Units; unit: Eyes] — Intravitreous anti-vascular endothelial growth factor drug that eye was receiving at time of enrollment.
  Eyes
    Aflibercept | 8
    Ranibizumab | 2
Prior injections with same anti-VEGF drug [Mean (Full Range); unit: Injections] — Number of injections with the same anti-VEGF drug prior to enrollment
  Injections | 21.9 [7 to 32]
Pseudophakic [Count of Units; unit: Eyes] — Number of eyes that had prior cataract surgery with an intraocular lens implant
  Eyes | 8
Current treatment interval [Count of Units; unit: Eyes] — Interval between intravitreal anti-VEGF injections prior to study enrollment. Same interval was maintained for study duration.
  Eyes
    Every 4 weeks | 8
    Every 5 weeks | 1
    Every 6 weeks | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Central Subfield Thickness (CST)
Description: Mean central subfield thickness (CST) on spectral domain optical coherence tomography (SD-OCT) on 1 visit prior to enrollment and all visits subsequent to study enrollment
Time Frame: 3 visits (8-12 weeks)
Population: Only 8 of 10 eyes completed study visit 3. The protocol only required follow-up through study visit 2.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Dorzolamide-timolol
Number analyzed (Participants) | 10
microns
  Pre-enrollment visit | 422.9 (100.9)
  Enrollment visit | 419.7 (95.9)
  Study visit 1 | 364.5 (76.3)
  Study visit 2 | 346.7 (99.9)
  Study visit 3: number analyzed (Participants) | 8
  Study visit 3 | 326.9 (115.5)
  Final visit | 334.1 (103.0)

2. Secondary Outcome: Visual Acuity
Description: LogMAR Visual acuity on enrollment and final visit
Time Frame: 3 visits (8-12 weeks)
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Dorzolamide-timolol
Number analyzed (Participants) | 10
Number analyzed (Eyes) | 10
logMAR
  Baseline | 0.54 (0.53)
  Final | 0.48 (0.29)

3. Secondary Outcome: Maximum Subretinal Fluid Height
Description: Measurement based on SD-OCT
Time Frame: 3 visits (8-12 weeks)
Population: Only 8 of 10 eyes completed study visit 3. The protocol only required follow-up through study visit 2.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Dorzolamide-timolol
Number analyzed (Participants) | 10
Number analyzed (Eyes) | 10
microns
  Pre-enrollment visit | 111.5 (101.3)
  Enrollment visit | 126.6 (78.2)
  Study visit 1 | 77.9 (70.7)
  Study visit 2 | 62.0 (59.7)
  Study visit 3: number analyzed (Participants) | 8
  Study visit 3: number analyzed (Eyes) | 8
  Study visit 3 | 56.5 (58.0)
  Final visit | 49.5 (54.1)

4. Secondary Outcome: Maximum Pigment Epithelial Detachment Height
Description: Measurement based on SD-OCT
Time Frame: 3 visits (8-12 weeks)
Population: Only 8 of 10 eyes completed study visit 3. The protocol only required follow-up through study visit 2.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Dorzolamide-timolol
Number analyzed (Participants) | 10
Number analyzed (Eyes) | 10
microns
  Pre-enrollment visit | 275.4 (170.7)
  Enrollment visit | 277.4 (174.9)
  Study visit 1 | 258.9 (173.7)
  Study visit 2 | 227.8 (163.0)
  Study visit 3: number analyzed (Participants) | 8
  Study visit 3: number analyzed (Eyes) | 8
  Study visit 3 | 275.4 (160.8)
  Final visit | 239.9 (163.0)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Dorzolamide-timolol
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No